CLINICAL TRIAL: NCT03143387
Title: Discomfort Evaluation During Atraumatic Restorative Treatment in Children- Clinical Trial
Brief Title: Discomfort Evaluation During Atraumatic Restorative Treatment in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty Sao Leopoldo Mandic Campinas (Other)
Responsible Party: Principal Investigator, Jose Carlos P Imparato, Principal Investigator, Faculty Sao Leopoldo Mandic Campinas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ART discomfort
Record Dates: First submitted 2017-02-21; First posted 2017-05-08 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Dental Caries; Primary Teeth; Post Dental Restoration
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atraumatic Restorative Treatment (Active Comparator): Partial removal of carious tissue using manual instruments.
  Interventions: Other: Caries removal using only manual instruments
- Chemo-mechanical Removal (Experimental): Partial removal of carious tissue using manual instruments and the material Chemo-mechanical removal group using Papacarie™gel.
  Interventions: Other: Caries removal using Papacarie gel

INTERVENTIONS:
Other: Caries removal using only manual instruments — Caries removal using only manual instruments according to Atraumatic Restorative Treatment
  Arms: Atraumatic Restorative Treatment
Other: Caries removal using Papacarie gel — Caries removal using a chemical-mechanical method - Papacarie gel and manual instruments.
  Arms: Chemo-mechanical Removal

SUMMARY:
This study evaluates the patient 's discomfort when submitted to partial caries removal through the atraumatic restorative treatment compared to chemo-mechanical caries removal using Papacarie™ gel.

DETAILED DESCRIPTION:
This study will evaluate the patient 's discomfort through oximeter (measuring the heart rate of the caries) prior to removal of the carious tissue, and when subjected to partial caries removal through the atraumatic restorative treatment compared to removal of chemo - mechanical caries with Papacarie gel ™.

ELIGIBILITY:
Inclusion Criteria:

* normoreactive,
* in good general health conditions,
* cooperative during screening,
* with at least one oclusal caries cavity in primary molars.
* Caregivers and/or children's parents must accept and sign the consent form.
* Children must accept their participation by nodding (assent).

Exclusion Criteria:

* pulp exposition,
* spontaneous pain,
* mobility,
* fistula,
* swollen area around the tooth,
* furcation,
* cervical lesion,
* restorations,
* sealants,
* developmental defect of enamel.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-10-15 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Discomfort evaluation with Wong-Baker | immediately after treatment
  The discomfort of each type of treatment will be evaluated using the facial scale of Wong-Baker (Wong, Baker, 1998).
  This scale indicates the discomfort of an individual who has to choose among six faces. The first image is a smiling happy face, indicating no discomfort, followed by gradually less cheerful expressions, up to the last one which is a very sad face covered by tears, indicating great discomfort. The participant will be asked to choose the face that is more similar to how he/she felt during the treatment immediately after the procedure. This answer should be given solely by the child, which means no parental or professional interference
Discomfort evaluation with heart beat and oxygen saturation | Before the procedure (when the patient is in the dental chair and there is no intervention), and during the procedure (removal of the cavity tissue).

SECONDARY OUTCOMES:
Time of restorative procedure | Will be evaluated the time required for removal of the caries tissue only with manual removal and when manual removal with the product Papacárie ™
Operators satisfaction | immediately after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Faculdade Sao Leopoldo Mandic, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berggren U, Meynert G. Dental fear and avoidance: causes, symptoms, and consequences. J Am Dent Assoc. 1984 Aug;109(2):247-51. doi: 10.14219/jada.archive.1984.0328. PMID 6590605
- [Background] Bussadori SK, Guedes CC, Bachiega JC, Santis TO, Motta LJ. Clinical and radiographic study of chemical-mechanical removal of caries using Papacarie: 24-month follow up. J Clin Pediatr Dent. 2011 Spring;35(3):251-4. doi: 10.17796/jcpd.35.3.75803m02524625h5. PMID 21678665
- [Background] Colares V, Franca C, Ferreira A, Amorim Filho HA, Oliveira MC. Dental anxiety and dental pain in 5- to 12-year-old children in Recife, Brazil. Eur Arch Paediatr Dent. 2013 Feb;14(1):15-9. doi: 10.1007/s40368-012-0001-8. Epub 2013 Jan 30. PMID 23532809
- [Background] Frencken JE, Holmgren CJ. Caries management through the Atraumatic Restorative Treatment (ART) approach and glass-ionomers: update 2013. Braz Oral Res. 2014;28:5-8. doi: 10.1590/S1806-83242013000600001. No abstract available. PMID 24402057
- [Background] Frencken JE, Leal SC, Navarro MF. Twenty-five-year atraumatic restorative treatment (ART) approach: a comprehensive overview. Clin Oral Investig. 2012 Oct;16(5):1337-46. doi: 10.1007/s00784-012-0783-4. Epub 2012 Jul 24. PMID 22824915
- [Background] Mattos-Silveira J, Floriano I, Ferreira FR, Vigano ME, Frizzo MA, Reyes A, Novaes TF, Moriyama CM, Raggio DP, Imparato JC, Mendes FM, Braga MM. New proposal of silver diamine fluoride use in arresting approximal caries: study protocol for a randomized controlled trial. Trials. 2014 Nov 19;15:448. doi: 10.1186/1745-6215-15-448. PMID 25409545
- [Background] Simon AK, Bhumika TV, Nair NS. Does atraumatic restorative treatment reduce dental anxiety in children? A systematic review and meta-analysis. Eur J Dent. 2015 Apr-Jun;9(2):304-309. doi: 10.4103/1305-7456.156841. PMID 26038668
- [Background] Staman NM, Townsend JA, Hagan JL. Observational study: discomfort following dental procedures for children. Pediatr Dent. 2013 Jan-Feb;35(1):52-4. PMID 23635899
- [Background] Soares FC, Lima RA, Santos Cda F, de Barros MV, Colares V. Predictors of dental anxiety in Brazilian 5-7years old children. Compr Psychiatry. 2016 May;67:46-53. doi: 10.1016/j.comppsych.2016.01.006. Epub 2016 Jan 21. PMID 27095334
- [Background] Venkataraghavan K, Kush A, Lakshminarayana C, Diwakar L, Ravikumar P, Patil S, Karthik S. Chemomechanical Caries Removal: A Review & Study of an Indigen-ously Developed Agent (Carie Care (TM) Gel) In Children. J Int Oral Health. 2013 Aug;5(4):84-90. Epub 2013 Aug 28. PMID 24155626